CLINICAL TRIAL: NCT04958889
Title: Symptoms and Biomarkers of Long COVID-19 in People Living With and Without HIV
Brief Title: COVID-19 Recovery Study: Symptoms and Biomarkers of Long COVID-19 in People Living With and Without HIV
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Rush University Medical Center (Other); University of California, San Francisco (Other); amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00278774
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV2); HIV
Keywords: COVID-19; Long COVID; HIV
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A mobile phlebotomist will draw blood at the participant's home at their convenience. The mobile phlebotomist will overnight ship blood samples using International Air Transport Association (IATA) approved procedures to the Immunology Specialty Lab at Rush University for processing, clinical laboratory testing, and storage. Work with samples will occur at Rush, Johns Hopkins and University of California, San Francisco (UCSF).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV+ adults with recent COVID-19 diagnosis: Required study visits:
  * Baseline questionnaire at enrollment or month 1.
  * Follow up questionnaire at month 1 and month 4
  * Height, weight, vital signs, and blood sampling at month 1 and month 4
  Optional study visits:
  • Follow up questionnaire at month 2, month 6, and month 12
  Interventions: Other: No intervention
- HIV- adults with recent COVID-19 diagnosis: Required study visits:
  * Baseline questionnaire at enrollment or month 1.
  * Follow up questionnaire at month 1 and month 4
  * Height, weight, vital signs, and blood sampling at month 1 and month 4
  Optional study visits:
  • Follow up questionnaire at month 2, month 6, and month 12
  Interventions: Other: No intervention
- HIV+ adults with no history of COVID-19: Required study visits:
  * Baseline questionnaire at enrollment.
  * Follow up questionnaire at enrollment and approximately 3 months after first follow up questionnaire.
  * Height, weight, vital signs, and blood sampling at enrollment.
  Optional study visits:
  • Follow up questionnaire at 1, 5, and 11 months after first follow up questionnaire.
  Interventions: Other: No intervention
- HIV- adults with no history of COVID-19: Required study visits:
  * Baseline questionnaire at enrollment.
  * Follow up questionnaire at enrollment and approximately 3 months after first follow up questionnaire.
  Optional study visits:
  • Follow up questionnaire at 1, 5, and 11 months after first follow up questionnaire.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — (observational study)

SUMMARY:
This observational study will prospectively characterize the long-term symptoms and side effects of COVID-19 in cohorts of people living with and without HIV. This will be achieved through a series of remote study visits involving completing surveys about health history, symptoms, mood, quality of life and changes in health, and up to two blood draws from home through the use of a mobile phlebotomy service.

DETAILED DESCRIPTION:
This is a prospective observational study being conducted to learn about late (2+ weeks or more) effects of COVID-19 in people living with and without HIV. The investigators plan to do this by studying people who have COVID-19 and people who have not had COVID-19, and by studying people living with HIV and people who are HIV-negative. The investigators will investigate the average duration of symptoms after COVID-19, how these symptoms affect quality of life, and what medical complications are common after COVID-19 in people with and without HIV.

Participation involves:

* Participant completion of surveys about themselves, their health history, their quality of life and mood in the recent past, and about COVID-19 or HIV if the participant has a history of either infection. The investigators will ask participants to answer questions in up to 5 follow-up surveys over the course of a year about their symptoms, mood, quality of life, and changes in health. Participants will also complete a series of short tests of thinking, memory, and reaction speed at certain follow-up surveys.
* Up to two visits to the participant's home (or an acceptable location of their choosing) by a phlebotomist. The phlebotomist will collect about 3.5 tablespoons of blood, as well as measure height, weight, and vital signs when laying down and standing up.

This is a fully remote study and all study activities can be done from home or another location of the participant's choosing.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Living within the contiguous 48 states
* Groups 1 and 3: self-reported HIV infection
* Groups 2 and 4: self-reported HIV negative

Exclusion Criteria:

* Inability to communicate by telephone in English or Spanish
* Inability to complete required study events
* A first or only diagnosis of COVID-19 5 or more weeks prior to first contact with participant
* Groups 3 and 4: diagnosis of cOVID-19 ever, or participant suspects they had COVID-19 at any time regardless of whether they were tested

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators will recruit volunteers with and without HIV and with and without a COVID-19 diagnosis from across the contiguous 48 US states in the following numbers:
  1. 110 adult people living with HIV (PWH) with COVID-19 symptom onset or first positive test within the prior 4 weeks
  2. 110 adult HIV-negative people with COVID-19 symptom onset or first positive test within the prior 4 weeks
  3. 45 adult PWH with no history of COVID-19
  4. 50 adult HIV-negative people with no history of COVID-19
  Investigators aim to enroll a population of PWH that is roughly representative of the demographic and geographic diversity of PWH across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity after COVID-19 infection over 12 months after infection | 1, 2, 4, 6 and 12 months
  Time to return to usual health and activities, as measured using the Influenza Patient-reported Outcome (Flu-PRO) instrument. The overall score is calculated as the mean across 32 items, and ranges from 0 (symptom free) to 4 (very severe symptoms).
Change in fatigue severity | 1 and 4 months
  Presence/absence of fatigue post-symptom onset, severity of fatigue and its effect on activity level as measured using the Fatigue Severity Scale. The Fatigue Severity Scale is a 9-item tool and each item is ranked from 1 (strongly disagree) to 7 (strongly agree). The item scores are added to generate the overall score, ranging from 9 (least severe) to 63 (most severe).
Change in number of COVID-19 symptoms experienced over 12 months after infection | 1, 2, 4, 6 and 12 months
  Number of symptoms experienced using Flu-PRO and additional COVID-19 specific symptoms in domains of neuropsychiatry, cardiovascular, and skin. Flu-PRO scores range from 0 (symptom free) to 4 (very severe symptoms).

SECONDARY OUTCOMES:
Change in mMRC rates of dyspnea | 1 and 4 months
  The Modified Medical Research Council (mMRC) instrument will be used to measure dyspnea. The mMRC rates severity of dyspnea on a scale of 0 to 4, 4 indicating the highest level of dyspnea severity.
Change in cognitive function (learning and memory) as measured by the RAVLT from month 1 to month 4 | 1 and 4 months
  Learning and memory assessed through the Rey Auditory Verbal Learning Test (RAVLT), in which participants receive a total learning score (range 0-36), a delayed recall score (range 0-12) and a recognition score (range -12 - +12). In all cases, a higher score indicates better recall.
Change in cognitive function (attention and executive function) as assessed through oral trail tests from month 1 to month 4 | 1 and 4 months
  Attention and executive function assessed through an oral trail test, in which participants are timed between 0 and 300 seconds. A higher time indicates lower attention and executive function.
Change in cognitive function (attention and working memory) as assessed through digit span tests from month 1 to month 4 | 1 and 4 months
  Attention and working memory assessed through a digit span task-forward and backward test. The forward test is scored from 0-16 and the backward test from 0-18, higher scores indicating better attention and memory.
Change in cognitive function (phonemic and semantic fluency) as assessed through letter and category-guided fluency tests from month 1 to month 4 | 1 and 4 months
  Phonemic and semantic fluency assessed through a letter-guided and category-guided fluency test. Scores range from 0-100, with a higher score indicating increased fluency.
Dysautonomia measured through orthostatic hypotension and orthostatic tachycardia | 1 month
  Orthostatic hypotension and orthostatic tachycardia (decrease in systolic blood pressure of 20 mmHg or decrease in diastolic blood pressure of 10 mmHg after 3 minutes of standing compared to sitting).
Dysautonomia measured through orthostatic hypotension and orthostatic tachycardia | 4 months
  Orthostatic hypotension and orthostatic tachycardia (decrease in systolic blood pressure of 20 mmHg or decrease in diastolic blood pressure of 10 mmHg after 3 minutes of standing compared to sitting).
Change in PHQ-9 depression symptoms | 1 and 4 months
  Self-reported measure of depressive symptoms using The Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9 item scale with a score range of 1-27 with higher scores indicating severe depression.
Change in quality of life as assessed using the Short Form-36 | 1 and 4 months
  Quality of life in the domains of vitality, physical functioning, bodily pain, general health perceptions, physical and emotional and social role functioning, as assessed using the Short Form-36. The Short Form-36 measures physical and mental health using 8 scales. The final score ranges from 0 (worse health status) to 100 (better health status).
Change in insomnia as assessed using the Insomnia Severity Index from month 1 to month 4 | 1 and 4 months
  Presence, severity, and patterns of insomnia, and its interference with daily functioning as assessed by the Insomnia Severity Index. The Insomnia Severity Index is a 7 item scale with a score range of 0-28. A higher score indicates severe insomnia.
Change in anxiety as assessed using the GAD-7 from month 1 to month 4 | 1 and 4 months
  Self-reported measure of anxiety using The Generalized Anxiety Disorder (GAD-7). The GAD-7 is a 7 item instrument used to measure or assess anxiety disorders. The score range is from 0-21. A higher score indicates severe anxiety.
Change in overall mental health as assessed using the CAT-MH from month 1 to month 4 | 1 and 4 months
  Self-reported measures of mental health symptoms (anxiety and depression) using the Computer Adaptive Test-Mental Health (CAT-MH). Scores range from 0-100, with a higher score indicating more severe symptoms.

OTHER OUTCOMES:
New self-reported diagnoses over 12 months after COVID-19 infection | 1, 2, 4, 6 and 12 months
  New medical diagnoses after COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Annie Antar, MD,PhD, Principal Investigator — Infectious Disease - Broadway
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No